CLINICAL TRIAL: NCT07306338
Title: Patient Interest in an Integrative Oncology Program at USC Norris Cancer Center: A Single-Institution Needs Assessment
Status: Not yet recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0S-25-3; NCI-2025-09248 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UP-25-00895; 0S-25-3 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2025-12-23; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients complete a survey and may participate in a focus group on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study

SUMMARY:
This study assesses patient perspectives on the interest in, feasibility, and acceptability of an Integrative Oncology Program for patients at USC NCCC and HC3 Women's Clinic.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To measure patient knowledge, attitudes, and interest in IO program services, identify predictors of willingness to participate or refer, and potential barriers to implementation into existing clinical care workflows.

OUTLINE: This is an observational study.

Patients complete a survey and may participate in a focus group on study.

ELIGIBILITY:
Inclusion Criteria:

* * Age ≥ 18 years

  * Ability to understand and the willingness to participate in the study.
  * English speaking
  * Patient of USC NCCC Outpatient Clinics or Keck HC3 Women's Health outpatient clinic.
  * Diagnosed solid or hematologic Malignancy

Exclusion Criteria:

* * Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid or hematologic cancer at USC NCCC outpatient clinics or Keck HC3 Women's Health outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Patient knowledge about Integrative Oncology (IO) program services | Through study completion, up to 1 year
  Outcome data will be collected through a survey per the study protocol. National Health Interview Survey (NHIS) - Complementary and Integrative Health (CDC 2024) module, Integrative Medicine Attitude Questionnaire (IMAQ) (Schneider, Meek, and Bell 2003), and Attitudes and Beliefs about Complementary and Alternative Medicines survey (Mao et al. 2012) will be used to quantify current use of and interest in integrative therapies for needs assessment.
Patient attitudes about IO program services | Through study completion, up to 1 year
  Outcome data will be collected through a survey per the study protocol. National Health Interview Survey (NHIS) - Complementary and Integrative Health (CDC 2024) module, Integrative Medicine Attitude Questionnaire (IMAQ) (Schneider, Meek, and Bell 2003), and Attitudes and Beliefs about Complementary and Alternative Medicines survey (Mao et al. 2012) will be used to quantify current use of and interest in integrative therapies for needs assessment.
Patient interest in IO program services | Through study completion, up to 1 year
  Outcome data will be collected through a survey per the study protocol. National Health Interview Survey (NHIS) - Complementary and Integrative Health (CDC 2024) module, Integrative Medicine Attitude Questionnaire (IMAQ) (Schneider, Meek, and Bell 2003), and Attitudes and Beliefs about Complementary and Alternative Medicines survey (Mao et al. 2012) will be used to quantify current use of and interest in integrative therapies for needs assessment.
Predictors of willingness to participate or refer | Through study completion, up to 1 year
  Outcome data will be collected through a survey per the study protocol. Adapted survey items from previously published studies (Larbi et al. 2021; Mao et al. 2014), including willingness to participate and pay will be used to asses this outcome.
Potential barriers to implementation | Through study completion, up to 1 year
  Outcome data will be collected through a survey per the study protocol. National Health Interview Survey (NHIS) - Complementary and Integrative Health (CDC 2024) module, Integrative Medicine Attitude Questionnaire (IMAQ) (Schneider, Meek, and Bell 2003), and Attitudes and Beliefs about Complementary and Alternative Medicines survey (Mao et al. 2012) will be used to quantify current use of and interest in integrative therapies for needs assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyue M Guo, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States